CLINICAL TRIAL: NCT01893892
Title: Double-blind, Randomized, Placebo-controlled Two-period Crossover Study to Assess the Effect of Levocarnitine on Vismodegib-associated Muscle Spasms
Brief Title: Levocarnitine in Treating Patients With Vismodegib-Associated Muscle Spasms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anne Chang, Associate Professor of Dermatology, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: SKIN0018; NCI-2013-01269 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 27478; P30CA124435 (NIH)
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Musculoskeletal Complications
Keywords: Basal Cell Carcinoma; Gorlin syndrome; Erivedge; Basal Cell Nevus Syndrome
MeSH Terms: conditions — Carcinoma, Basal Cell; Basal Cell Nevus Syndrome | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (levocarnitine start) (Experimental): Patients receive levocarnitine PO BID during weeks 1-4. Washout is weeks 5-8. Patients then cross-over to placebo for weeks 9-12.
  Interventions: Dietary Supplement: levocarnitine; Other: questionnaire administration
- Arm II (placebo start) (Placebo Comparator): Patients receive placebo PO BID during weeks 1-4. Washout is weeks 5-8. Patients then cross-over to levocarnitine for weeks 9-12.
  Interventions: Other: placebo; Other: questionnaire administration

INTERVENTIONS:
Dietary Supplement: levocarnitine — Given PO
  Other Names: Carnitor; L-carnitine
  Arms: Arm I (levocarnitine start)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo start)
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies levocarnitine in treating patients with vismodegib-associated muscle spasms. Levocarnitine may decrease muscle spasms caused by vismodegib.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of levocarnitine on muscle spasm frequency compared to placebo (median percentage comparison)

SECONDARY OBJECTIVES:

I. To assess intensity of muscle spasms after levocarnitine compared to placebo.

II. To assess responses related to activities of daily living or psychosocial function after levocarnitine compared to placebo.

III. To assess the number of body locations affected by muscle spasms after levocarnitine or placebo.

IV. To assess the frequency and severity of all adverse effects on levocarnitine versus placebo.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive levocarnitine orally (PO) twice daily (BID) during weeks 1-4. Washout is from weeks 5-8. Patients then cross-over to placebo PO twice daipy for weeks 9-12.

ARM II: Patients receive placebo PO twice daily during weeks 1-4. Washout is from weeks 5-8. Patients then cross-over to levocarnitine for weeks 9-12.

ELIGIBILITY:
Inclusion Criteria:

* Taking vismodegib daily
* Subject answers item #1 of muscle spasms questionnaire as moderate or severe intensity at time of screening
* At least one muscle spasm per day at time of screening
* Muscle spasms onset after starting vismodegib
* Willing and able to understand and sign consent form

Exclusion Criteria:

* Presence of muscle spasms or active neurologic disease prior to start of vismodegib
* Use of thyroid medication at the time of screening
* Use of Coumadin or acenocoumarol at time of screening
* Change in regimen of muscle relaxant medications within four weeks of enrollment
* If on stable muscle relaxant medication regimen for 4 weeks prior to enrolling, not willing to maintain muscle relaxant regimen without change during course of the study
* Presence of significant renal disease or hemodialysis which would result in dramatic reductions of systemic levocarnitine levels
* History of seizures
* Known deficiency in carnitine (genetic, etc.)
* Any uncontrolled medical condition which may place the patient at increased risk during study participation (at the discretion of the clinical investigator)
* Unable or unwilling to comply with study procedures
* Pregnant or lactating
* All female patients of childbearing potential including those who are within 1 year of last menstrual period will be required to take a pregnancy test during screening, enrollment and at week 0, 4, 8 and 12
* If female of reproductive age, or male partner of female of reproductive age, unwilling to use two medically reliable forms of birth control while on vismodegib
* Unwilling to refrain from donation of bodily fluid (blood, platelets, etc.) within 7 months of last vismodegib dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Percentage difference in muscle spasm frequency (defined as number per week) between levocarnitine and placebo | 12 weeks
  Wilcoxon rank-sum test, paired

SECONDARY OUTCOMES:
Change in severity of muscle spasms after levocarnitine and placebo | 12 weeks
  Wilcoxon rank-sum test, paired
Change in number of body locations affected by muscle spasms after levocarnitine and placebo | 12 weeks
  Wilcoxon rank-sum test, paired
Change in impact of spasms on activities of daily living (such as sleeping or driving) after levocarnitine and placebo | 12 weeks
  as measured on questionnaire items
Social/emotional impacts of muscle spasms after levocarnitine and placebo | 12 weeks
  as measured on questionnaire items
Frequency of adverse events after levocarnitine and placebo | 12 weeks
  according to CTCAE 4.03
Severity of adverse events after levocarnitine and placebo | 12 weeks
  according to CTCAE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lynn Chang, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States